CLINICAL TRIAL: NCT01198665
Title: A Phase I/II Study of RAD001 Combined With CHOP in Newly Diagnosed Peripheral T-cell Lymphomas
Brief Title: RAD001 Combined With CHOP in Newly Diagnosed Peripheral T-cell Lymphomas
Acronym: RADCHOP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Yonsei University (Other); National Cancer Center, Korea (Other Government); Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Associate professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01-001
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral T Cell Lymphoma Unspecified; Anaplastic Large Cell Lymphoma, ALK-negative; Angioimmunoblastic T Cell Lymphoma; Cutaneous T Cell Lymphoma
Keywords: RAD001; chemotherpy; T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous | interventions — Everolimus; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001-CHOP (Experimental): Prospective multicenter open-label phase I/II study Phase I: RAD001 2.5 - 10 mg PO daily D1-14 + CHOP every 3 weeks Phase II: Determined dosage of RAD001 + CHOP every 3 weeks Treatment will be continued until planned 6 cycles or disease progression
  Interventions: Drug: RAD001 (Everolimus)

INTERVENTIONS:
Drug: RAD001 (Everolimus) — Phase I Level 1: RAD001 2.5 mg PO daily D1-14 + CHOP Level 2: RAD001 5 mg PO daily D1-14 + CHOP Level 3: RAD001 7.5 mg PO daily D1-14 + CHOP Level 4: RAD001 10 mg PO daily D1-14 + CHOP CHOP every 3 weeks D1 Cytoxan 750mg/m2 + D5W 100ml MIV over 1hr D1 Doxorubicin 50mg/m2 + D5W 100ml MIV over 30mins D1 Vincristine 1.4mg/m2 (max.2mg) IV push D1-D5 Prednisolone 100mg/d PO (40-30-30) Phase II Determined dosage of RAD001 + CHOP every 3 weeks
  Other Names: Cytoxan, Doxorubicin, Vincristine, prednisolone

SUMMARY:
The urgent need for new effective therapy for T-cell lymphoma patients and promising results observed so far in trials with RAD001(everolimus, mTOR inhibitor) strongly warrants the investigation of RAD001 combined with CHOP as a first-line treatment in peripheral T-cell lymphoma patients.

Thus, we designed a phase I/II study with the combination of RAD001 with CHOP chemotherapy for newly diagnosed peripheral T-cell lymphoma patients.

Phase I

1. Primary objective

   : To define the maximum tolerable dose
2. Secondary objective

   * To evaluate the dose-limiting toxicity
   * To evaluate the pharmacokinetics of RAD001
   * Pharmacogenomic profiling

Phase II

1. Primary objective

   : To evaluate the overall response rate
2. Secondary objective

   * To estimate the time to progression
   * To estimate overall survival
   * Pharmacogenomic profiling

DETAILED DESCRIPTION:
Phase I Level 1: RAD001 2.5 mg PO daily D1-14 + CHOP Level 2: RAD001 5 mg PO daily D1-14 + CHOP Level 3: RAD001 7.5 mg PO daily D1-14 + CHOP Level 4: RAD001 10 mg PO daily D1-14 + CHOP CHOP every 3 weeks D1 Cytoxan 750mg/m2 + D5W 100ml MIV over 1hr D1 Doxorubicin 50mg/m2 + D5W 100ml MIV over 30mins D1 Vincristine 1.4mg/m2 (max.2mg) IV push D1-D5 Prednisolone 100mg/d PO (40-30-30) Phase II Determined dosage of RAD001 + CHOP every 3 weeks Treatment will be continued until planned 6 cycles or disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven peripheral T-cell lymphoma, unspecified, (PTCL), ALK-negative anaplastic large cell T-cell lymphoma (ALCL), Angioimmunoblastic T cell lymphoma (AITL), Cutaneous T-cell lymphoma
2. Adequate organ function as defined by the following criteria:

   A.Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy B.Total serum bilirubin ≤1.5 x ULN C.Absolute neutrophil count (ANC) ≥1500/µL D.Platelets ≥100,000/µL E.Hemoglobin ≥9.0 g/dL (may be transfused or erythropoietin treated) F.Serum calcium ≤12.0 mg/dL G.Serum creatinine ≤1.5 x ULN
3. At least one measurable lesion
4. ECOG PS 0-2
5. Informed consent
6. Age 20 to 70 years old

Exclusion Criteria:

1. Prior radiation therapy or surgery within 4 weeks prior to study entry
2. History of central nervous system (CNS) metastases
3. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
4. Pregnancy or breastfeeding.
5. Hepatitis B virus surface antigen positive
6. Extranodal NK/T cell lymphoma
7. Mycosis fungoides
8. ALK-positive Anaplastic large cell lymphoma

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
determination of the maximum tolerable dose and evaluation of response rate | Phase I for maximal tolerable dose and phase II for efficacy

SECONDARY OUTCOMES:
doe-limiting toxicity and pharmacogenomics | Phase I/II
  Phase I
  * To evaluate the dose-limiting toxicity
  * To evaluate the pharmacokinetics of RAD001
  * Pharmacogenomic profiling Phase II
  * To estimate the time to progression
  * To estimate overall survival
  * Pharmacogenomic profiling

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - National Cancer Center, Goyang-si, Kyoungki-do
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Yonsei Medical Center, Severance Hospital, Seoul